CLINICAL TRIAL: NCT00521885
Title: Arixtra(Fondaparinux) vs. Lovenox (Enoxaparin) in Prevention of DVT in Acute Medically Ill, Non-surgical Patients
Brief Title: Comparison of Arixtra vs. Lovenox to Prevent Blood Clots in Medically Ill Patients
Acronym: BRiEF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped due to lack of accrual
Sponsor: Lehigh Valley Hospital (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LVH IRB# 2-20070508
Record Dates: First submitted 2007-08-24; First posted 2007-08-28 (Estimated); Results first posted 2017-11-01 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2017-11

CONDITIONS: Venous Thrombosis
Keywords: Bleeding rates; Prophylaxis for deep vein thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — Fondaparinux; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arixtra (Fondaparinox) 2.5 mg SC Daily (Active Comparator): Arixtra (Fondaparinox) 2.5 mg SC Daily
  Interventions: Drug: Arixtra (Fondaparinox) 2.5 mg SC Daily
- Lovenox 40mg SC Daily (Active Comparator): Lovenox 40mg SC Daily
  Interventions: Drug: Lovenox 40mg SC Daily

INTERVENTIONS:
Drug: Arixtra (Fondaparinox) 2.5 mg SC Daily — Patients will be randomized to receive Arixtra 2.5mg once a day if randomized to this arm
  Other Names: fondaparinux
  Arms: Arixtra (Fondaparinox) 2.5 mg SC Daily
Drug: Lovenox 40mg SC Daily — Patients will be randomized to receive Lovenox 40mg SC Daily if randomized to this arm
  Other Names: enoxaparin
  Arms: Lovenox 40mg SC Daily

SUMMARY:
A total of 50 patients >40 yrs of age with an expected hospital stay in the Medical Intensive Care or Regional Heart Unit at LVH Muhlenberg of 6 days or longer will be enrolled. The patient and study team will be blinded to which drug they are receiving (either Arixtra or Lovenox). Subjects will be examined for any bleeding complications. Subjects will receive drug for a total of 6-14 days while in the hospital. A follow up phone call will be performed by the study team approximately 30 days after discharge from the hospital.

DETAILED DESCRIPTION:
A total of 50 patients will be enrolled in this double-blinded, randomized, controlled trial. Inclusion criteria: subjects>40 yrs of age with an expected hospital stay in the Medical Intensive Care or Regional Heart Unit at LVH Muhlenberg of 6 days or longer (4 days bedridden) will be enrolled. Total drug treatment will be 6-14 days while in the hospital. A follow up phone call will be performed by the study team approximately 30 days after hospital discharge. Primary endpoint: bleeding rate (minor vs major) between study days 1-14. Secondary endpoint: DVT study days 1-14 (confirmed with LE duplex ultrasonogram).

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 40 years of age.
* Pt with expected stay in hospital 6 days or >, with expectation to be bedridden for > 4 days.
* Pts admitted to the MICU, Regional Heart Units of LV-MHC

Exclusion Criteria:

* Surgical primary admission diagnosis
* Recent surgery within the past 12 weeks
* Planned surgery on the current admission
* Pregnancy
* Vent-dependent respiratory failure requiring intubation for >24 hours.
* Known current DVT or PE prior to enrollment in study.
* Creatinine clearance < 30 mL/min (calculated by the Cockcroft-Gault method) in a well-hydrated patient.
* Hx of prior or current lower upper or lower GI bleed.
* Platelet count < 100,000 per cubic millimeter
* Current or prior anticoagulation within the prior 48 hours, excluding a single dose &lor 24 hour period of prophylactic agent
* Bacterial endocarditis.
* Hemophilia
* Hypersensitivity to aspirin.
* Hypersensitivity to Arixtra or Lovenox
* Hx of hemorrhagic or ischemic stroke < 3 months prior to enrolling
* Hematocrit < 28%.
* SBP >200 mmHg or DBP >120 mmHg
* Positive for occult blood in stool.
* Admission to hospital for > 48 hours prior to randomization
* Documented congenital or acquired bleeding disorder
* Indwelling intrathecal or epidural catheter
* Life expectancy < 30 days
* Inability to have a flu assessment post-discharge from the hospital

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kruklitis, MD, Principal Investigator — Lehigh Valley Hospital
Locations (1):
- Lehigh Valley Hospital Muhlenberg, Bethlehem, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Unable to recruit suitable subjects is the reason this study was terminated early
Pre-assignment Details: one patient was a screened failure- after consent found to have an exclusion criteria during screening
Groups:
- Arixtra (Fondaparinox) 2.5 mg Given Subcutaneously (SC) Daily: In this arm subjects will be randomized to Arixtra (Fondaparinox) 2.5 mg given Subcutaneously (SC) once a day starting on day 1 and continuing through day 14 or day of discharge, whichever comes first.
  Arixtra: Arixtra 2.5mg Sc Daily
- Lovenox 40mg Subcutaneously (SC) Daily: Subjects will be randomized using a random generated listing of numbers with arm assignments associated with each assigned number. Only the study pharmacist will have access to this randomization code. All other study team members will remain blinded to the treatment arm. In this arm subjects will be randomized to Lovenox 40mg Subcutaneously (SC) Daily starting on day 1 and continuing through day 14 or day of discharge, whichever comes first.
  Lovenox: Lovenox 40mg SC Daily
Period: Overall Study
Arm/Group | Arixtra (Fondaparinox) 2.5 mg Given Subcutaneously (SC) Daily | Lovenox 40mg Subcutaneously (SC) Daily
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: see comments under "limitations"- the study apparently enrolled 1 participant and it is not documented which group that patient was assigned to- so we cannot confirm patients in either group- the total enrolled is 1. The study was done so long ago no one from the study team is available and there is no documentation as to which group this 1 patient was randomized to.
Groups:
- Arixtra (Fondaparinox) 2.5 mg Given SubCutaneously Daily: Subjects may be randomized to Arixtra (Fondaparinox) 2.5 mg given SubCutaneously Daily starting on day 1 and continuing through day 14 or day of discharge, whichever comes first
  Arixtra: Arixtra 2.5mg Sc Daily
- Lovenox 40mg SubCutaneously Daily: Subjects may be randomized to Lovenox 40mg SubCutaneously Daily starting on day 1 and continuing through day 14 or day of discharge, whichever comes first
  Lovenox: Lovenox 40mg SC Daily
- Total: Total of all reporting groups
Arm/Group | Arixtra (Fondaparinox) 2.5 mg Given SubCutaneously Daily | Lovenox 40mg SubCutaneously Daily | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Bleeding Rate Study Day 1-14 (Minor vs Major) With 30 Day f/u
Description: Bleeding Rate- Major bleeding defined as one or a combination of the following: Fatal; Bleeding at critical organ sites (intracranial, retroperitoneal, intraocular, pericardial, spinal or adrenal). Minor Bleeding defined as clinically overt bleeding that is not major bleeding.
Time Frame: 14 days
Population: There was only 1 patient enrolled and it is not documented anywhere which group they were assigned to- the study is so old and no one is here who would know; therefore I cannot verify any patients in either group
Groups:
- Arixtra (Fondaparinox) 2.5 mg Given Subcutaneously (SC)Once a: Arixtra (Fondaparinox) 2.5 mg given Subcutaneously (SC)once a day
  Arixtra: Arixtra 2.5mg Sc Daily
- Lovenox 40mg Subcutaneously (SC) Daily: Lovenox 40mg Subcutaneously (SC) Daily
  Lovenox: Lovenox 40mg SC Daily
Arm/Group | Arixtra (Fondaparinox) 2.5 mg Given Subcutaneously (SC)Once a | Lovenox 40mg Subcutaneously (SC) Daily
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Deep Vein Thrombosis
Description: Confirmed by Lower Extremity Ultra-sonogram
Time Frame: 14 Days
Population: There was 1 patient enrolled and it is not documented which group the patient was assigned therefore I cannot verify which group the patient should be included.
Arm/Group | Arixtra (Fondaparinox) 2.5 mg Given Subcutaneously (SC)Once a | Lovenox 40mg Subcutaneously (SC) Daily
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 14 days
Description: Does not differ
Groups:
- Arixtra (Fondaparinox) 2.5 mg Given SC Daily: Arixtra (Fondaparinox) 2.5 mg given Subcutaneously (SC)once a day
  Arixtra: Arixtra 2.5mg Sc Daily
- Lovenox 40mg SC Daily: Lovenox 40mg Subcutaneously (SC) Daily
  Lovenox: Lovenox 40mg SC Daily
Arm/Group | Arixtra (Fondaparinox) 2.5 mg Given SC Daily | Lovenox 40mg SC Daily
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Began 2007 and ended 2009-1 subject enrolled-no SAE noted. No records which arm enrolled subject was assigned, so cannot accurately fill the patient flow section as "1" to match enroll number. Unknown what arm subject in. Only blinded pharm.was aware

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes